CLINICAL TRIAL: NCT05833191
Title: Efficacy of Different Nerve Stimulation Methods in Individuals With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chronic Constipation
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Constipation
Keywords: vagus; tibial nerve stimülation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The study will be included in a 12-session treatment program over four weeks.
Who Masked: Investigator
Masking Description: In our study, which is planned as a single-blind evaluation, different physiotherapists will perform the evaluation and application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular vagus stimulation (Experimental): Non-invasive transcutaneous devices stimulate the vagus nerve via the auricular route or from the carotid.
  Interventions: Device: Auricular vagus stimulation
- Tibial Nerve Stimulation (Experimental): Transcutaneous tibial nerve stimulation (TTNS) is reported to be beneficial for fecal and urinary incontinence. A review of the literature showed that there are very few studies using TTNS that have been shown to be effective for constipation.
  Interventions: Device: Tibial Nerve Stimulation

INTERVENTIONS:
Device: Auricular vagus stimulation — When the nervus tibialis approaches the medial malleolus, it approaches the surface. In this study, bilateral transcutaneous electrical nerve stimulation (TENS) electrodes will be placed under the medial malleolus approximately at the point where the tibialis nerve contacts the surface.
  Arms: Auricular vagus stimulation
Device: Tibial Nerve Stimulation — When the nervus tibialis approaches the medial malleolus, it approaches the surface. In this study, bilateral transcutaneous electrical nerve stimulation (TENS) electrodes will be placed under the medial malleolus approximately at the point where the tibialis nerve contacts the surface.
  Arms: Tibial Nerve Stimulation

SUMMARY:
Constipation is the most common digestive complaint in the general population. Normal stool frequency ranges from at least three times a week to a maximum of two times a day. Constipation can be classified into three main groups as constipation with normal transit time, constipation with slow transit time and dyssynergic defecation disorders.

DETAILED DESCRIPTION:
In chronic constipation, treatment should be directed towards the underlying cause. In the treatment of chronic constipation, lifestyle changes and physiotherapy are in the first place, pharmacological treatment is in the second place, and surgical treatment is in the third place. Physiotherapy modalities such as defecation training, classical massage, electrical stimulation, anorectal biofeedback and exercise training can be used in the treatment of chronic constipation.

ELIGIBILITY:
Inclusion criteria:

•Being diagnosed with chronic constipation

Exclusion criteria:

* Metabolic diseases
* Severe heart or kidney disease, previous gastrointestinal, spinal or pelvic surgery other than cholecystectomy, hysterectomy or appendectomy,
* Neurological diseases such as multiple sclerosis, stroke, Parkinson's disease or spinal injury, impaired awareness
* Mini-mental score < 15
* Legal blindness, pregnancy, rectal prolapse, anal fissure, and alternating pattern of constipation and diarrhea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Scale | 4 weeks
  Bristol Stool Scale (BGS) In the scale, the type of stool is classified into 7 different groups. In the Bristol stool scale, the intestinal transit time of stool is evaluated over seven different stool types. According to BGS, 1-2 points are "hard stools", 3-4-5 points are "normal stools" and 6-7 points are "soft-watery stools (diarrhea)".
Pelvic Pain Impact Questionnaire | 4 weeks
  The clinical assessment of the effect of pelvic pain on women consists of 10 questions. However, the first 8 questions are scored. The range of points to be taken from the questionnaire varies between 1 and 32. As the score to be obtained from the questionnaire increases, the degree of functional limitation of pelvic pain on the person also increases.
Superficial Electromyography Biofeedback | 4 weeks
  Before starting the treatment, the target that the patient wants to reach is determined. With the "set target" feature on the device, tensing and relaxation are practiced for 10 seconds and the average target is determined. Then, the target is created by taking the percentage of this determined target. Since the goal in this study is relaxation, the patient is asked to decrease the value on the graph during the session.
Constipation Severity Scale | 4 weeks
  The lowest possible total score is 0, and the highest is 73. A high score from the scale indicates that the symptoms are serious. The highest score that can be obtained from the five-point Likert-type scale is 140, and the lowest score is 28. It is thought that as the scores obtained from the scale increase, the quality of life is negatively affected.
Autonomic nervous system device | 4 weeks
  In the study, the autonomic nervous system will be evaluated with the Polar H10 device. By connecting the device to a smart phone via bluetooth, the data will be recorded and the software supported by the device will be used for the analysis of the data. A measurement will be made with the participant in a sitting position and lasting up to 3 minutes.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Medipol hospital, Istanbul, Istanbul Avrupa Kitasi
  - Medipol hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan K, Wells CI, Dinning P, Bissett IP, O'Grady G. Placebo Response Rates in Electrical Nerve Stimulation Trials for Fecal Incontinence and Constipation: A Systematic Review and Meta-Analysis. Neuromodulation. 2020 Dec;23(8):1108-1116. doi: 10.1111/ner.13092. Epub 2019 Dec 30. PMID 31889364